CLINICAL TRIAL: NCT03512444
Title: Does Circumferential Negative Pressure Therapy Impair Distal O2 Saturation? A Randomized Controlled Study
Brief Title: Does Circumferential Negative Pressure Therapy Impair Distal O2 Saturation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Aljomah (Other)
Responsible Party: Sponsor-Investigator, Ahmed Aljomah, Research Associate, King Faisal Specialist Hospital & Research Center
Organization: King Faisal Specialist Hospital & Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2181026
Record Dates: First submitted 2018-04-09; First posted 2018-04-30 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Negative Pressure Wound Therapy; Wound
Keywords: negative pressure therapy; negative pressure; Wound therapy; NPWT; Vacuum therapy; VAC
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: 2 groups: intervention and control (both are in each arm of the same participant).
  Intervention will be applied at one arm (chosen randomly) with using the contralateral arm as a control.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative pressure (Experimental): Negative pressure system is applied with negative pressure (Active)
  at a participant's unilateral arm
  Interventions: Device: Negative Pressure System
- No negative pressure (No Intervention): Negative pressure system is applied without negative pressure (Inactive)
  at a participant's contralateral arm

INTERVENTIONS:
Device: Negative Pressure System — Negative Pressure System is a non-invasive system that applies sub-atmospheric(Negative) pressure, through a foam and an air-tight film dressing which is connected by suction tubes to a controller unit by which the primary negative pressure can be adjusted.
  Arms: Negative pressure

SUMMARY:
Abstract:

Background: Circumferential negative pressure wound therapy (CNPWT) is commonly used to manage wounds and enhance the healing process. A theoretical concern was recently raised that CNPWT may have a negative effect on perfusion distally. Objectives: We aim to evaluate the effect of circumferential negative pressure therapy (CNPT) on distal O2 saturation in healthy volunteers. Design: Randomized controlled non-inferiority study. Methods: Fourteen healthy adult volunteers with O2 saturation ≥95% (by index finger pulse oximetry) will be invited to participate in the study. After obtaining a written informed consent, CNPWT foam/dressing will be applied in a sandwich-like manner on the middle third of each arm and a negative intermittent pressure of 125 mmHg will be applied to one arm chosen randomly, using the contralateral arm as control. The pressure will be applied 5 minutes on and 2 minutes off for 9 hours. Individual's participation will be terminated if O2 saturation drops below 92% at any study time. The outcome measure is index finger O2 saturation and will be checked every 30 minutes using a pulse oximetry. The area under the curve (AUC) of O2 saturation in the 2 arms will be compared using ANCOVA. Sample size was calculated to have 90% power, assuming a type one error of 5%, non-inferiority margin of 24 (mean AUC difference), SD of 20, and drop out of 2 participants. Importance: The study is expected to provide conclusive evidence on the effect of intermittent CNPT on distal O2 saturation. The results would have direct implications for CNPWT.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of circumferential negative pressure therapy (CNPT) on distal O2 saturation in healthy volunteers.

Design and Methodology:

Design: This is a randomized controlled non-inferiority study.

Recruitment: Volunteers will be recruited through advertisement in King Faisal Specialist Hospital & Research Centre and other hospitals in Riyadh.

Pre-study procedures: After obtaining a well documented medical history each volunteer will undergo a full physical examination as well as an in-depth upper limb examination and comprehensive evaluation (including a pre-study index finger O2 saturation and upper limbs circumference measurements), the following data will be also collected: age, sex, height&weight, body mass index, and vital signs.

Procedures: CNPWT foam and dressing (in accordance to manufacturer's instructions) will be applied in a sandwich-like manner on the middle third of each arm, and a negative intermittent pressure of 125 mmHg will be applied to one arm chosen randomly, using the contralateral arm as control. The pressure will be applied 5 minutes on and 2 minutes off for 9 hours. Individual's participation will be terminated if O2 saturation by pulse oximetry drops below 92% at any study time.

Statistical analysis: The area under the curve (AUC) of O2 saturation will be compared between the 2 arms using ANCOVA.

Randomization schedule: a randomization schedule will be generated by an online program (www.randomization.com). Block randomization will be used.

Sample size: Fourteen adult volunteers will be invited to participate in the study.

The sample size for the study was calculated to have 90% power, assuming a type one error of 5%, non-inferiority margin of 24 (mean AUC difference), SD of 20, and drop out of 2 participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers with O2 saturation ≥95% by pulse oximetry. Potential volunteers will be screened by routine medical history and physical examination and an in-depth upper limb examination

Exclusion Criteria:

* Unhealthy individual
* Chronic conditions
* History of upper limb diseases or defects.
* History of upper limb Surgical intervention.
* History of upper limb implants.
* Pre-study O2 saturation in either indices of less than 95%
* Congenital or Traumatic upper limb defect

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of index finger O2 saturation over 9 hours. | 9 hours
  Index finger O2 saturation will be checked every 30 minutes using a pulse oximetry, from zero hour of the study until the end of the 9th hour, then AUC will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PHD, Principal Investigator — King Faisal Specialist Hospital & Research Center; Ahmed S Aljomah, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: open access after publication

REFERENCES:
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Morykwas MJ, Faler BJ, Pearce DJ, Argenta LC. Effects of varying levels of subatmospheric pressure on the rate of granulation tissue formation in experimental wounds in swine. Ann Plast Surg. 2001 Nov;47(5):547-51. doi: 10.1097/00000637-200111000-00013. PMID 11716268
- [Background] Vikatmaa P, Juutilainen V, Kuukasjarvi P, Malmivaara A. Negative pressure wound therapy: a systematic review on effectiveness and safety. Eur J Vasc Endovasc Surg. 2008 Oct;36(4):438-48. doi: 10.1016/j.ejvs.2008.06.010. Epub 2008 Aug 3. PMID 18675559
- [Background] Ubbink DT, Westerbos SJ, Nelson EA, Vermeulen H. A systematic review of topical negative pressure therapy for acute and chronic wounds. Br J Surg. 2008 Jun;95(6):685-92. doi: 10.1002/bjs.6238. PMID 18446777
- [Background] Kairinos N, Solomons M, Hudson DA. Negative-pressure wound therapy I: the paradox of negative-pressure wound therapy. Plast Reconstr Surg. 2009 Feb;123(2):589-598. doi: 10.1097/PRS.0b013e3181956551. PMID 19182617
- [Background] Kairinos N, Voogd AM, Botha PH, Kotze T, Kahn D, Hudson DA, Solomons M. Negative-pressure wound therapy II: negative-pressure wound therapy and increased perfusion. Just an illusion? Plast Reconstr Surg. 2009 Feb;123(2):601-612. doi: 10.1097/PRS.0b013e318196b97b. PMID 19182619
- [Background] Othman D. Negative pressure wound therapy literature review of efficacy, cost effectiveness, and impact on patients' quality of life in chronic wound management and its implementation in the United kingdom. Plast Surg Int. 2012;2012:374398. doi: 10.1155/2012/374398. Epub 2012 May 30. PMID 22701169
- [Background] Moues CM, Heule F, Hovius SE. A review of topical negative pressure therapy in wound healing: sufficient evidence? Am J Surg. 2011 Apr;201(4):544-56. doi: 10.1016/j.amjsurg.2010.04.029. PMID 21421104